CLINICAL TRIAL: NCT04296162
Title: A Phase II Study to Assess the Effectiveness and Safety of Oral Vinorelbine or Capecitabine Combined With Trastuzumab as Adjuvant Treatment for Patients With Lymph Node Negative, HER-2 Positive and Small Tumor Size Breast Cancer (ORCHID)
Brief Title: Oral Vinorelbine or Capecitabine Combined With Trastuzumab as Adjuvant Treatment for Patients With Lymph Node Negative, HER-2 Positive and Small Tumor Size Breast Cancer (ORCHID)
Acronym: ORCHID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1503144-7
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: oral vinorelbine; capecitabine; trastuzumab; adjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): 6 cycle of oral vinorelbine or capecitabine combined with trastuzumab (21 days per cycle), followed by sequential single trastuzumab to 1 year
  Interventions: Drug: Vinorelbine; Drug: Capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine chemotherapy (oral)
Drug: Capecitabine — Capecitabine chemotherapy (oral)
Drug: Trastuzumab — Trastuzumab target therapy

SUMMARY:
This is a prospective, open-lable Phase II clinical trial (ORCHID study) evaluating the effectiveness and safety of oral vinorelbine or capecitabine combined with trastuzumab as adjuvant treatment for patients with lymph node negative, HER-2 positive and small tumor size breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. women aged 18-70 years old;
2. T ≤1cm and negative lymph node confirmed by histopathology after early breast cancer surgery
3. HER2 positive confirmed by histopathology after early breast cancer surgery（HER2-positive breast cancer defined as a positive in situ hybridization test or an Immunohistochemistry (IHC) status of 3+. If IHC is 2+, a negative in situ hybridization (Fluorescence in situ hybridization (FISH), Chromogenic in situ hybridization (CISH) , or Silver in situ hybridization (SISH)) test is required by local laboratory testing.)
4. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN，and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula).
6. Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy）;
2. Has bilateral breast cancer;
3. Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
4. Has metastic (Stage 4) breast cancer;
5. Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
6. Patients participating in other clinical trials at the same time;
7. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
8. Has severe or uncontrolled infection;
9. Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
10. the researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 year

SECONDARY OUTCOMES:
distant disease free survival | 5 year
overall survival | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhi-Ming Shao, Shanghai, China